CLINICAL TRIAL: NCT02314598
Title: Therapy Coil Electrogram Collection Study
Acronym: TEC
Status: Terminated | Type: Observational
Why Stopped: No chance to meet the foreseen target of patients with study endpoint
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Other Study IDs: TEC Study
Record Dates: First submitted 2014-10-30; First posted 2014-12-11 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Lead Insulation Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment

SUMMARY:
This is a prospective, non-randomized, multicenter, post market release study which will collect electrograms (EGMs) from patients at risk of a suspected insulation failure to the high voltage portion of the defibrillator lead and will evaluate the electrogram signals.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign and date the study Informed Consent form
* Subject is at least 18 years of age (or older, if required by local law)
* Subject is willing and able to wear a Holter monitor for up to 24 hours
* Subject has been implanted with a Medtronic ICD or CRT-D device
* Subject has an increased risk of lead insulation breach

Exclusion Criteria:

* Subject has medical conditions that would limit study participation
* Subject is enrolled in one or more concurrent studies that would confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an Implantable Cardioverter Defibrillator (ICD) or a Cardiac Resynchronization Therapy Defibrillator (CRT-D) device followed-up at community hospitals
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Slovakia (2):
  - SUSCCH, Banská Bystrica
  - NUSCH, Bratislava

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Patients at risk of suspected insulation failure to the high voltage portion of the defibrillator lead
Period: Overall Study
Arm/Group | All Study Participants
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Slovakia | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Abnormal Electrograms During a Lead Issue
Description: Number of patients with at least one instance of abnormal noise during recording. Electrograms will be collected during 24 hours and afterwards abnormalities in the electrograms will be visually identified.
Time Frame: 24 hours
Population: 46 subjects were enrolled and completed the study. All subjects met the inclusion and exclusion criteria.
  5 subjects were excluded since they did not have an Holter recording with at least 12 hours of telemetry.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 41
Participants | 0

2. Secondary Outcome: Proportion of Patients With Abnormal Electrograms and Lead Failure
Description: Compare the proportion of patients with abnormal electrograms (e.g. high frequency spike) and a high voltage lead failure within 1 month to those patients with abnormal electrograms and no lead failure within 1 month
Time Frame: 1 month
Population: There were no patients with a high voltage lead failure, therefore the proportions cannot be estimated nor compared.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Additional Abnormal Electrogram Characteristics
Description: Identify additional characteristics in the Far-field Electrograms that may halp to identify patients at risk of a high voltage lead failure
Time Frame: 1 month
Population: There were no patients with a high voltage lead failure, therefore the additional characteristics cannot be identified.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: No adverse event collected in this study
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
41 out of the 46 enrolled subjects completed a Holter recording with at least 12 hours of telemetry, but none of them reached any study endpoint.

Therefore enrollment and study were closed and foreseen analyses could have not been performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-08-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT02314598/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT02314598/SAP_001.pdf